CLINICAL TRIAL: NCT01604486
Title: Natural Ischaemic Preconditioning Before First Myocardial Infarction: an Analysis of Prospectively Collected UK Electronic Primary Care Records Linked to the National Registry of Acute Coronary Syndromes
Brief Title: Natural Ischaemic Preconditioning Before First Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Emily Herrett, Research Degree Student, London School of Hygiene and Tropical Medicine
Other Study IDs: EH CALIBER IP; 086091/Z/08/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Myocardial Infarction; Angina Pectoris; Coronary Heart Disease; Peripheral Arterial Disease; Cerebrovascular Disease
Keywords: Myocardial infarction; Ischaemic preconditioning; Myocardial Ischaemia National Audit Project; General Practice Research Database; Hospital Episode Statistics; Office for National Statistics
MeSH Terms: conditions — Myocardial Infarction; Angina Pectoris; Coronary Disease; Peripheral Arterial Disease; Cerebrovascular Disorders

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- MI without ischaemic preconditioning: Myocardial infarction unheralded by any previous cardiovascular disease diagnosis and without symptoms of chest pain in the previous 90 days.
- MI with longstanding disease: Patients with myocardial infarction who have had diagnosed atherosclerotic disease for longer than 90 days preceding infarct.
- MI with only chest pain: Patients with chest pain in the 90 days preceding MI, but with no prior atherosclerotic disease diagnoses.
- MI with disease and chest pain: Myocardial infarction occurring with previously diagnosed atherosclerotic disease of longer than 90 days' duration, but with chest pain in 90 days preceding infarct.

SUMMARY:
There is a sharp rise in the rate of coronary heart disease diagnoses and chest pain consultations in the 90 days before a first heart attack. There is some evidence that chest pain and angina symptoms in this period have a beneficial effect on heart attack outcomes in hospital and shortly after discharge. However, the available evidence is lacking in three key areas. First it is based on a retrospective patient report of symptoms after the heart attack has occurred; this means that patients are required to survive their heart attack and may make errors when reporting prior symptoms. Second, evidence for an effect on longer term outcomes, and coronary outcomes in particular (e.g. coronary death, further heart attacks) are unknown. Third, there is conflicting evidence that these effects might differ by age, in men and women, and according to treatment in hospital.

The investigators hope to address the limitations in the evidence by performing a large, prospective study of the occurrence, timing and effect of different types of symptoms and disease diagnoses occurring before heart attack.

The investigators hypothesise that prospectively collected, clinical measures of chest pain symptoms and cardiovascular diagnoses in primary care will have a beneficial effect on short term coronary mortality and may have a beneficial effect on longer term coronary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients in GPRD practices which are deemed "up to standard" by GPRD criteria will be included if their practice agreed to be linked to the MINAP, HES and ONS datasets.
* Patients must have at least one year of GPRD "up to standard" registration before the date of first MI.
* Age over 18.
* First myocardial infarction occurring between 1st January 2003 and 31st December 2008, as recorded in the Hospital Episode Statistics data or the Myocardial Ischaemia National Audit Project.

Exclusion Criteria:

* Patients will be excluded if they do not fulfil one of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of patients with a first myocardial infarction who are registered at those GPRD practices that agreed to the linkage with the MINAP database, and whose practices are "up to standard" according to GPRD criteria. Practices taking part in the GPRD are chosen to be representative of all UK practices, and 98% of people in the UK are registered with a GP. Therefore the GPRD should be a representative sample of the UK population.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Recurrent myocardial infarction | Up to seven years
  Myocardial infarction occurring thirty or more days after the study start date.

SECONDARY OUTCOMES:
Coronary mortality | Up to seven years
  Coronary mortality, using ONS mortality statistics (ICD-10 codes I20-I25)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Herrett, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Harry Hemingway, FRCP, Study Director — University College, London
Locations (1):
- London School of Hygiene and Tropical Medicine, London, United Kingdom

REFERENCES:
- [Derived] Herrett E, Bhaskaran K, Timmis A, Denaxas S, Hemingway H, Smeeth L. Association between clinical presentations before myocardial infarction and coronary mortality: a prospective population-based study using linked electronic records. Eur Heart J. 2014 Sep 14;35(35):2363-71. doi: 10.1093/eurheartj/ehu286. Epub 2014 Jul 19. PMID 25038774